CLINICAL TRIAL: NCT02310789
Title: (Study: Vertex IIS) A Study To Access the Effects of Ivacaftor on Wild Type CFTR-Open Probability (PO) In The Sweat Gland Secretory Coil
Brief Title: (Study: Vertex IIS) Does Ivacaftor Alter Wild Type CFTR-Open Probability In The Sweat Gland Secretory Coil?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Barry Moss (Other)
Responsible Party: Sponsor-Investigator, Richard Barry Moss, Professor of Pediatrics at the Lucile Salter Packard Children's Hospital, Emeritus, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 31238
Record Dates: First submitted 2014-09-03; First posted 2014-12-08 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ivacaftor (Experimental): Participants will receive ivacaftor orally for 3 days, followed by 35 days off drug. Participants will repeat this cycle then receive ivacaftor for 3 additional days. For sweat testing, participants will receive β-adrenergic cocktail to stimulated sweating, at both 1% stimulation strength and full stimulation strength. Each participant will also receive pilocarpine nitrate 5% administered by Macroduct sweat stimulator device. Sweat stimulation testing will be done on- and off-ivacaftor.
  Interventions: Drug: Ivacaftor; Drug: β-Adrenergic cocktail; Drug: Pilocarpine Nitrate 5%; Device: Macroduct sweat stimulator

INTERVENTIONS:
Drug: Ivacaftor — 150mg administered orally twice daily.
  Other Names: Kalydeco
Drug: β-Adrenergic cocktail — Administered subcutaneously to induce sweating. Cocktail composed of atropine (280µM), isoproterenol (160µM), and aminophylline (20 mM).
Drug: Pilocarpine Nitrate 5% — Administered subcutaneously using Macroduct sweat stimulator device.
Device: Macroduct sweat stimulator

SUMMARY:
Clinical studies of lumacaftor + ivacaftor (combo therapy) produced better FEV1 (forced expiratory volume in 1 second) improvements than ivacaftor alone, without further improvement in sweat chloride results.

To help understand why sweat chloride was unresponsive, the investigators will use a newly developed sweat secretion test that provides accurate, in vivo readout of CFTR (cystic fibrosis transmembrane conductance regulator) function in the sweat gland secretory coil.

The investigators devised a protocol to determine if short courses of ivacaftor (3.5 days) will produce significant increases in WT (Wild-Type, i.e. normal) CFTR open probability by measuring CFTR-dependent sweating (C-sweat) in subjects with WT CFTR.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disease caused by malfunctioning of a protein called CFTR.

CF affects various organs including the sweat glands and the lungs. An FDA approved drug called ivacaftor helps some people with CF, and laboratory tests show that it produces further improvement when combined with an investigational drug called lumacaftor. However, results from clinical tests of the two drugs used together gave mixed results: lung function improved but sweat gland function did not improve. This study will measure CFTR-dependent sweat rate to test the hypothesis that CFTR in the normal sweat glands might be functioning at peak efficiency, and so can't be improved further with ivacaftor, thus accounting for the apparent discrepancy between lung function and sweat gland results. CFTR-dependent sweat rate is important to understanding CF because it is a very accurate measure of CFTR function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults without a Cystic Fibrosis (CF) mutation
* Carriers with a known CF mutation

Exclusion Criteria:

1. Documented liver disease
2. Participants should not be taking:

   * medicines that are strong CYP3A (Cytochrome P450, family 3, subfamily A) inducers, such as:

     * the antibiotics rifampin and rifabutin;
     * seizure medications (phenobarbital, carbamazepine, or phenytoin); and
     * the herbal supplement St. John's Wort, substantially decreases exposure of ivacaftor and may diminish effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wine, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

REFERENCES:
- See also: Sweat rate analysis of ivacaftor potentiation of CFTR in non-CF adults — https://www.nature.com/articles/s41598-018-34308-8

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivacaftor: Participants received ivacaftor orally for 3 days, followed by 35 days off drug. Participants repeated this cycle then received ivacaftor for 3 additional days. For sweat testing, participants received β-adrenergic cocktail to stimulated sweating, at both 1% stimulation strength and full stimulation strength. Each participant also received pilocarpine nitrate 5% administered by Macroduct sweat stimulator device. Sweat stimulation testing was done on- and off-ivacaftor.
Period: Overall Study
Arm/Group | Ivacaftor
Started | 8
Completed | 7
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ivacaftor
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 46.5 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Healthy Volunteers [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Cystic Fibrosis Transmembrane Conductance Regulator (CFTR)-Dependent Sweat Rate
Description: CFTR-dependent sweat rate (C-sweat) was analyzed using a linear mixed model, combining on- and off-ivacaftor data.
Time Frame: Up to 79 days
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ivacaftor
Number analyzed (Participants) | 7
percent change
  1% β-adrenergic stimulation | 16.45 (2.25)
  Full β-adrenergic stimulation | 6.60 (2.97)

2. Secondary Outcome: Change Sweat Chloride Production
Description: Sweat chloride concentration was measured via the traditional sweat collection methods using the pilocarpine stimulation with the Macroduct device.
Time Frame: Up to 79 days
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ivacaftor
Number analyzed (Participants) | 7
percent change
  On ivacaftor | 25.1 (11.4)
  Off Ivacaftor | 24.9 (6.1)

ADVERSE EVENTS:
Time Frame: Up to 79 days
Arm/Group | Ivacaftor
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor (N=8)
Subcutaneous induration (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes